CLINICAL TRIAL: NCT02561754
Title: Weight Management for Adolescents With IDD
Acronym: IDDAdol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001857; 5R01HD079642 (NIH)
Record Dates: First submitted 2015-06-25; First posted 2015-09-28 (Estimated); Results first posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Developmental Disabilities; Weight Loss; Body Weight; Down Syndrome; Body Weight Changes; Intellectual Disability
Keywords: Diet; Obesity; Adolescents; Intellectual and Developmental Disability
MeSH Terms: conditions — Developmental Disabilities; Weight Loss; Body Weight; Down Syndrome; Body Weight Changes; Intellectual Disability; Obesity | interventions — Technology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Face-To-Face/CD (Active Comparator): Delivery: Face-to-face Diet: Conventional diet
  Interventions: Dietary Supplement: Conventional Diet (CD); Behavioral: Face-to-face (FTF)
- Technology delivery/CD (Experimental): Delivery: Technology Diet: Conventional diet
  Interventions: Dietary Supplement: Conventional Diet (CD); Behavioral: Technology (TECH); Other: iPad with FaceTime
- Technology delivery/eSLD (Experimental): Delivery: Technology Diet: enhanced Stop Light Diet
  Interventions: Dietary Supplement: Enhanced Stop Light Diet (eSLD); Behavioral: Technology (TECH); Other: iPad with FaceTime

INTERVENTIONS:
Dietary Supplement: Enhanced Stop Light Diet (eSLD) — eSDL includes reduced energy portion controlled meals for 6 months, encouraged consumption of lower energy shakes and 35 fruits and vegetables per week.
  Arms: Technology delivery/eSLD
Dietary Supplement: Conventional Diet (CD) — CD is a nutritionally balanced, reduced energy, high volume, lower fat ( fat=20-30% energy) diet.
  Arms: Face-To-Face/CD; Technology delivery/CD
Behavioral: Face-to-face (FTF) — FTF will meet with a health educator in person and will track progress using pen and paper records for both physical activity and diet.
  Arms: Face-To-Face/CD
Behavioral: Technology (TECH) — TECH groups will receive the intervention using an iPad with the FaceTimeTM application for video meetings with a health educator and will track progress using the Lose it! application for both physical activity and diet.
  Arms: Technology delivery/CD; Technology delivery/eSLD
Other: iPad with FaceTime — TECH groups will receive the intervention using an iPad with the FaceTimeTM to the intervention field.
  Arms: Technology delivery/CD; Technology delivery/eSLD

SUMMARY:
The goal of this study is to explore the impact of two different diets (conventional vs. enhanced stop light) and two different delivery systems (face-to-face vs. remote) on weight across 18 months in overweight and obese adolescents with intellectual and developmental disabilities.

DETAILED DESCRIPTION:
Rates of obesity and obesity related chronic health conditions are higher in adolescents with Intellectual and Developmental Disabilities (IDD) than those in the general population. Many of the negative health consequences observed in obese adults are already present in obese adolescents with IDD.

This study is a 3 group randomized trial to evaluate the intervention delivery system and type of reduced energy diet. The investigators will randomize 123 overweight/obese adolescents with mild to moderate IDD to one of 3 groups for an 18 month trial (6 month weight loss; 12 month weight maintenance):

group 1) Face-To-Face/CD

group 2) Technology delivery/CD

group 3) Technology delivery/eSLD.

All participants will receive a progressive program of physical activity. Participants on the CD diet will be asked to consume a nutritionally balanced, reduced energy, high volume, lower fat ( fat=20-30% energy) diet. Participants on the eSLD will consume pre-packaged portion controlled meals with the addition of 5 fruits and vegetables per day.

FTF will meet with a health educator and will track progress using pen and paper records for both physical activity and diet. TECH groups will receive the intervention using an iPad with the FaceTimeTM application for video meetings with a health educator and will track progress using the Lose it! application for both physical activity and diet.

ELIGIBILITY:
Inclusion Criteria:

* Age 13-21 yrs
* Mild (IQ of 74-50) or moderate (IQ 40-49) IDD,
* Of sufficient functional ability to understand directions, communicate preferences (e.g. foods), wants (e.g. more to eat/drink), and needs (e.g. assistance with food preparation) through spoken language.
* Overweight or obese (BMI ≥ 85th%ile on CDC growth charts, or waist circumference to height ratio > 0.5
* Living at home with a parent or guardian.
* Internet access in the home.
* No plans to relocate outside the study area over the next 18 mos
* Physician consent for PA and diet.

Exclusion Criteria:

* Insulin dependent diabetes
* Participation in a weight management program involving diet and PA in the past 6 mos
* Eating disorders, serious food allergies, consuming special diets, aversion to common foods,
* Diagnosis of Prader-Willi Syndrome
* Currently pregnant, planning on/becoming pregnant during the study.
* Unable to participate in moderate to vigorous PA.

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 110 (Actual)
Dates: Start 2015-03; Primary Completion 2020-05-12 (Actual); Study Completion 2021-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph E Donnelly, EdD, Principal Investigator — University of Kansas Medical Center
Locations (2):
- United States (2):
  - University of Kansas Medical Center, Kansas City, Kansas
  - Energy Balance Lab, The University of Kansas, Lawrence, Kansas

REFERENCES:
- [Derived] Bodde AE, White DA, Forseth B, Hastert M, Washburn R, Donnelly J, Sullivan D, Ptomey LT. Parent factors associated with BMI, diet, and physical activity of adolescents with intellectual and developmental disabilities. Disabil Health J. 2023 Oct;16(4):101507. doi: 10.1016/j.dhjo.2023.101507. Epub 2023 Jul 7. PMID 37487764
- [Derived] Bodde AE, Helsel BC, Hastert M, Suire KB, Washburn RA, Donnelly JE, Ptomey LT. The prevalence of obesity and lifestyle behaviors of parents of youth with intellectual and developmental disabilities. Disabil Health J. 2023 Jul;16(3):101430. doi: 10.1016/j.dhjo.2022.101430. Epub 2022 Dec 14. PMID 36604240
- [Derived] Ptomey LT, Lee J, White DA, Helsel BC, Washburn RA, Donnelly JE. Changes in physical activity across a 6-month weight loss intervention in adolescents with intellectual and developmental disabilities. J Intellect Disabil Res. 2022 Jun;66(6):545-557. doi: 10.1111/jir.12909. Epub 2021 Dec 16. PMID 34915594
- [Derived] Ptomey LT, Washburn RA, Goetz JR, Sullivan DK, Gibson CA, Mayo MS, Krebill R, Gorczyca AM, Montgomery RN, Honas JJ, Helsel BC, Donnelly JE. Weight Loss Interventions for Adolescents With Intellectual Disabilities: An RCT. Pediatrics. 2021 Sep;148(3):e2021050261. doi: 10.1542/peds.2021-050261. Epub 2021 Aug 19. PMID 34413247

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Face-To-Face/CD | Technology Delivery/CD | Technology Delivery/eSLD
Started | 36 | 39 | 35
6 Months | 35 | 39 | 30
12 Months | 32 | 34 | 26
Completed | 30 | 33 | 26
Not Completed | 6 | 6 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Face-To-Face/CD | Technology Delivery/CD | Technology Delivery/eSLD | Total
Number analyzed (Participants) | 36 | 39 | 35 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.3 (2.7) | 15.6 (1.7) | 16.7 (2.5) | 16.2 (2.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 24 | 18 | 58
  Male | 20 | 15 | 17 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4 | 8
  Not Hispanic or Latino | 34 | 37 | 31 | 102
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 4 | 7
  White | 30 | 38 | 29 | 97
  More than one race | 3 | 1 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 88.4 (29.5) | 74.9 (16.5) | 83.6 (26.4) | 81.9 (26.3)

OUTCOME MEASURES:

1. Primary Outcome: Weight Change at 6 Months
Description: Participants will be weighed in shorts and a t-shirt , on a calibrated scale to the nearest 0.1 kg.
Time Frame: Change in weight from baseline to 6 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Face-To-Face/CD | Technology Delivery/CD | Technology Delivery/eSLD
Number analyzed (Participants) | 35 | 39 | 30
kg | -0.3 (5.0) | -1.8 (4.0) | -5.0 (5.9)

2. Secondary Outcome: Weight Change Across 18 Months
Description: Participants will be weighed in shorts and a t-shirt between 7 and 10 AM, in duplicate, on a calibrated scale to the nearest 0.1 kg.
Time Frame: Change in weight from baseline to 18 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Face-To-Face/CD | Technology Delivery/CD | Technology Delivery/eSLD
Number analyzed (Participants) | 30 | 33 | 26
kg | 1.4 (9.7) | -0.2 (6.6) | -2.2 (7.4)

ADVERSE EVENTS:
Time Frame: Across 18 months
Arm/Group | Face-To-Face/CD | Technology Delivery/CD | Technology Delivery/eSLD
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/39 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/39 | 1/35
Other Adverse Events (participants affected / at risk) | 0/36 | 5/39 | 1/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Face-To-Face/CD (N=36) | Technology Delivery/CD (N=39) | Technology Delivery/eSLD (N=35)
Open Heart Surgery (Surgical and medical procedures) | NA | NA | 1 (1) — Durning study participant discovered they had a congenital heart defect and required surgery to repair. Need for surgery was unrelated to the intervention
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Face-To-Face/CD (N=36) | Technology Delivery/CD (N=39) | Technology Delivery/eSLD (N=35)
Broken Bone (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1
Colonoscopy (Surgical and medical procedures) | 0 | 1 | 0
Pericardial Effusion (Cardiac disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-30): https://cdn.clinicaltrials.gov/large-docs/54/NCT02561754/Prot_SAP_000.pdf